CLINICAL TRIAL: NCT06026852
Title: Validation of Uncertainty Quantifying Machine Learning Models to Predict Beta-lactam Antimicrobial Concentrations in ICU Patients
Brief Title: Validation of Betalactam ML Prediction Models - TDMAide
Acronym: TDMAide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Research Foundation Flanders (Other); Imec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIV-23-04-042892
Record Dates: First submitted 2023-06-09; First posted 2023-09-07 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Infections
Keywords: Artificial Intelligence; Machine Learning; PK/PD; Piperacillin-tazobactam; Meropenem; Intensive Care Unit
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Other): Patients admitted to the ICU who are treated with piperacillin-tazobactam or meropenem.
  Interventions: Device: Prediction of plasma concentration of piperacillin-tazobactam or meropenem; Diagnostic Test: Determination of plasma concentration of piperacillin-tazobactam or meropenem
- Physicians (Other): Physicians in training or consultants who care for patients that are included in the study.
  Interventions: Other: Daily short questionnaire

INTERVENTIONS:
Device: Prediction of plasma concentration of piperacillin-tazobactam or meropenem — For included patients, a prediction will be made by developed machine learning models about the expected plasma concentration of piperacillin-tazobactam or meropenem by using routinely collected health care data.
  Arms: Patients
Diagnostic Test: Determination of plasma concentration of piperacillin-tazobactam or meropenem — For included patients, the total plasma concentration of piperacillin-tazobactam or meropenem will be determined. Were possible, this will be done using a blood sample that was collected during routine daily bloodwork which is performed in the morning. If no routine sample is available, a study specific sample will be drawn at approximately the same time as a routine sample would be drawn.
  Arms: Patients
Other: Daily short questionnaire — Physicians who care for patients included in the study will be asked to fill in a short daily questionnaire that evaluates the perceived necessity and added value of daily therapeutic drug monitoring.
  Arms: Physicians

SUMMARY:
The goal of this study is to learn about the real wold behavior of developed machine learning models that predict the plasma concentration of piperacillin-tazobactam and meropenem in critically ill patients admitted to the intensive care unit (ICU).

The main aim of the study is to validate the performance of these machine learning models. To this end, daily measured plasma concentrations of the investigated antimicrobials will be compared with the predicted concentration by the machine learning algorithms.

Additional goals of the study include:

* To describe the total plasma concentration over time of piperacillin-tazobactam and meropenem in patients admitted to the ICU.
* To quantify the correlation between plasma concentrations of piperacillin-tazobactam and meropenem and the development of side effects.
* To evaluate the perceived necessity of therapeutic drug monitoring (TDM) of consultants and physicians in training working in the ICU.
* To evaluate the perceived added value of daily TDM.

Samples (where possible taken routinely) from participating patients will be analyzed for meropenem and piperacillin-tazobactam plasma concentration. Participating physicians will be asked to fill in a short daily questionnaire during the time a patient under their care is treated with the antimicrobial under investigation.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Admission to the ICU.
* Age above 18 years old.
* Treatment with piperacillin-tazobactam or meropenem for less than 48 hours.

Exclusion Criteria:

* Pregnant or lactating patients.
* Limitation of therapy beyond "Do not resuscitate".
* Expected demise within 48 hours after inclusion.
* Haemoglobin < 7 g/dL.
* Previous inclusion in this study for a treatment course with the same antimicrobial.

Consultants and physicians in training

Inclusion Criteria:

* Consultant or physician in training working in the ICU.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-09-26 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Difference between predicted (TDMAIde) and measured (via HPLC-MS/MS method) plasma concentrations | Through study completion, an average of 1 year
  The difference between the predicted concentration (from the TDMAide software) and the concentration range based on the measured concentration (measured from the blood sample from the patient and analyzed using a HPLC-MS/MS method, with and without taking into account intra- and inter measurement variabilities of the HPLC-MS/MS method.

SECONDARY OUTCOMES:
Plasma concentration (determined via HPLC-MS/MS) trends | Through study completion, an average of 1 year
  Trends in total plasma concentration over time of piperacillin-tazobactam and meropenem in patients admitted to the ICU
Correlation between plasma concentrations (measured by HPLC-MS/MS) and side effects as percentage of patients experiencing the side effect | Through study completion, an average of 1 year
  The correlation between plasma concentrations of piperacillin-tazobactam and meropenem and the development of renal (decline in urinary output, rise in serum creatinin), gastro-intestinal (C. difficile infections, stool consistency, elevation of ALT/AST/gamma GT/Alkalic fosfatase/INR/APTT/bilirubin), neurological (delirium as measured by Intensice Care Delirium Screening Checklist - ICDSC) or hematological (Rise or fall of thrombocytes, development of leucopenia/agranulocytosis/eosinophelia/hemolytic anemia) side effects.
Perceived necessity of therapeutic drug monitoring | Through study completion, an average of 1 year
  The perceived necessity of therapeutic drug monitoring of consultants and physicians in training working in the ICU by evaluating the perceived necessity collected during the surveys with the measured plasma concentrations.
Perceived added value of therapeutic drug monitoring | Through study completion, an average of 1 year
  The perceived added value of daily therapeutic drug monitoring from the responses to the survey

CONTACTS AND LOCATIONS:
Overall Officials: Jan De Waele, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available upon reasonable request and after approval by the appropriate ethical and regulatory bodies.
Supporting Information: ICF, CSR, Analytic Code
Time Frame: At publication of the results
Access Criteria: Individual participant data will be made available upon reasonable request and after approval by the appropriate ethical and regulatory bodies.